CLINICAL TRIAL: NCT01765179
Title: Phase III, Open-label Study of the Safety and Efficacy of Oral Testosterone Undecanoate (TU)in Hypogonadal Men
Brief Title: Safety and Efficacy Trial of Testosterone Undecanoate
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Clarus Therapeutics, Inc. (Industry)
Collaborators: inVentiv Health Clinical (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLAR-12011
Record Dates: First submitted 2013-01-08; First posted 2013-01-10 (Estimated); Results first posted 2017-09-21 (Actual); Last update posted 2017-12-12 (Actual); Status verified 2017-11

CONDITIONS: Male Hypogonadism
Keywords: testosterone; male hypogonadism; low testosterone
MeSH Terms: conditions — Eunuchism | interventions — testosterone undecanoate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Oral testosterone undecanoate (Experimental)
  Interventions: Drug: Oral testosterone undecanoate

INTERVENTIONS:
Drug: Oral testosterone undecanoate — Initial dose 200 mg T, BID; dose titration Days 42 and/or 84 based on serum T levels obtained 3-5 hours post AM dose on Days 30 and 72. Dosages increased or decreased in 50 mg increments.

SUMMARY:
The purpose of the study is to determine if oral testosterone undecanoate is effective and safe in the treatment of low testosterone in men.

ELIGIBILITY:
Inclusion Criteria:

* Serum testosterone of less than or equal to 300 ng/dL (the mean of two samples collected 1 hour apart in the morning between 6:00 and 10:00 AM)

Exclusion Criteria:

* Significant intercurrent disease of any type, in particular liver, kidney, uncontrolled or poorly controlled heart disease including hypertension, CHF or CAD, or psychiatric illness including depression.
* Recent history of stroke, including transient ischemic attack (TIA) or acute coronary event
* Untreated, severe obstructive sleep apnea
* Hematocrit <35% or >48%
* Serum transaminases >2 times upper limit of normal, serum bilirubin >2.0 mg/dL, and serum creatinine >2.0 mg/dL
* BMI > or equal to 38
* Stable doses of lipid-lowering medication for less than three months
* Stable doses of oral medication for diabetes for less than two months
* Abnormal prostate digital rectal examination [palpable nodule(s)], elevated PSA (serum PSA >3.9 ng/mL), IPSS score > or equal to 19 points, and /or history of prostate cancer.
* History of breast cancer
* Use of dietary supplement saw palmetto or phytoestrogens and use of any dietary supplements that may increase serum T, such as androstenedione or DHEA with the previous 4 weeks
* Know malabsorption syndrome and/or current treatment iwht oral lipase inhibitors
* Known history of abuse of alcohol or any drug substance with the previous 2 years
* Current use of antiandrogens, estrogens, oral CYP3A4 inducers or inhibitors, or long-acting opioid analgesics
* Receipt of any drug as part of a research study within 30 days of initial dose administration in this study
* Blood donation within the 12 week period before initial dose administration in this study

Ages: 18 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Actual)
Dates: Start 2013-01; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ronald Swerdloff, MD, Principal Investigator — Los Andgeles Biomedical Research Institute
Locations (27):
- United States (27):
  - Alabama Clinical Therapeutics, LLC, Birmingham, Alabama
  - Alabama Internal Medicine, PC, Birmingham, Alabama
  - Medical Affliated Research Center, Inc., Huntsville, Alabama
  - Precision Trials/Valley Urologic Associates, Glendale, Arizona
  - Premier Clinical Research Center, Phoenix, Arizona
  - Precision Trials/Valley Urologic Associates, Phoenix, Arizona
  - Quality of LIfe Medical and Research Center, Tucson, Arizona
  - SC Clinical Research, Inc., Garden Grove, California
  - South ORange County Endocrinology, Laguna Hill, California
  - Tower Urology, Tower Research Institute, Los Angeles, California
  - San Diego Sexual Medicine, San Diego, California
  - LABiomedical Research Institute at Harbor-UCLA Medical Center, Torrance, California
  - Conneticut Clinical Research Center, Middlebury, Connecticut
  - South Florida Medical Research, Aventura, Florida
  - PAB Clinical Research, Brandon, Florida
  - Innovative Research of West Florida, Clearwater, Florida
  - Jacksonville Impotence Treatment Center, Jacksonville, Florida
  - University Urology Associates, New York, New York
  - Sunstone Medical Research, Medford, Oregon
  - Unrologic Consultants of SE Pennsylvania, Bala-Cynwyd, Pennsylvania
  - Research Across America, Carrollton, Texas
  - Research Across America, Dallas, Texas
  - Clinical Trial Network, Houston, Texas
  - Potenium Clinical Research, LLC, Hurst, Texas
  - Clinical Trials of Texas, Inc., San Antonio, Texas
  - Rainer Clinical Research Center, Inc., Renton, Washington
  - University of Washington, Seattle, Washington

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Oral Testosterone Undecanoate
Started | 144
Completed | 117
Not Completed | 27
Not completed — Adverse Event | 3
Not completed — Lost to Follow-up | 5
Not completed — Non-compliance with study drug | 2
Not completed — Protocol Violation | 1
Not completed — Withdrawal by Subject | 8
Not completed — Hematocrit >54% | 3
Not completed — prohibited med | 1
Not completed — Out of country unable to finish study | 1
Not completed — lack of venous access | 1
Not completed — work conflict | 1
Not completed — Ca elevated 10.6 | 1

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set
Arm/Group | Oral Testosterone Undecanoate
Number analyzed (Participants) | 144
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 116
  >=65 years | 28
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.8 (10.60)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 144
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: American Indian or Alaskan Native | 1
  Race: Asian | 13
  Race: Black or African American | 15
  Race: Native Hawaiian or Other Pacific Islander | 0
  Race: White | 114
  Race: Other | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 144

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Treated Patients With an Average Serum Testosterone (T) Concentration (Cavg) Between 300 and 1000 ng/dL
Description: The number of subjects (116) analyzed includes only those subjects with serum testosterone Cavg data available on study day 114.
Time Frame: 0, 1, 2, 3, 4, 6, 8, 12, 24, 48, 72, 96 hours post-dose on day 114
Population: The number of subjects (116) analyzed includes only those subjects with serum testosterone Cavg data available on study day 114.
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Testosterone Undecanoate
Number analyzed (Participants) | 116
Participants | 87

2. Secondary Outcome: Percentage of Treated Patients With Maximum Serum T Concentrations (Cmax) Values in Selected Ranges on Day 114 Efficacy Population
Description: as for outcome 1
Time Frame: 0, 1, 2, 3, 4, 6, 8, 12, 24, 48, 72, 96 hours post-dose on day 114
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Testosterone Undecanoate
Number analyzed (Participants) | 116
Participants
  Cmax less that 1500 ng/dL | 95
  Cmax between 1500 and 1800 ng/dL | 10
  Cmax >1800 to 2500 ng/dL | 7
  Cmax >2500 ng/dL | 4

ADVERSE EVENTS:
Arm/Group | Oral Testosterone Undecanoate
All-Cause Mortality (participants affected / at risk) | 0/144
Serious Adverse Events (participants affected / at risk) | 2/144
Other Adverse Events (participants affected / at risk) | 46/144
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Oral Testosterone Undecanoate (N=144)
Cerebrovascular accident (Nervous system disorders) | 1 (1) — Moderate stroke considered definitely not related by investigator
chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) — exacerbation of COPD considered definitely not related by investigator
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Oral Testosterone Undecanoate (N=144)
diarrhea (Gastrointestinal disorders) | 5
dyspepsia (Gastrointestinal disorders) | 4
eructation (Gastrointestinal disorders) | 3
haemorrhoids (Gastrointestinal disorders) | 3
oedema peripheral (General disorders) | 4
nasopharyngitis (Infections and infestations) | 3
upper respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 5
blood creatinine increased (Investigations) | 3
blood glucose increased (Investigations) | 3
haematocrit (Investigations) | 3
gout (Metabolism and nutrition disorders) | 3
prostatomegaly (Reproductive system and breast disorders) | 3
hypertension (Vascular disorders) | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days